CLINICAL TRIAL: NCT00490204
Title: A Randomized, Double Blind, Placebo Controlled Study for Evaluation of the Efficacy and Safety of Cetirizine Dry Syrup (CTZ DS) (2.5 mg or 5 mg Twice a Day) in Children (2 Years of Age or Older But Under 15 Years Old) Suffering From Perennial Allergic Rhinitis.
Brief Title: Cetirizine Placebo Controlled Study For Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 110458
Record Dates: First submitted 2007-06-19; First posted 2007-06-22 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial Allergic Rhinitis; Placebo control; anti-histamine; Cetirizine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetirizine

SUMMARY:
Study objective is to verify the superiority of CTZ DS to the placebo groups in the change of total nasal symptom score (TNSS) over the total treatment period from the score of the baseline assessment period.

ELIGIBILITY:
Inclusion criteria:

- [Before the start of observation period]

1. Children with a history of hypersensitivity to an ingredient of cetirizine hydrochloride preparation, or hydroxyzine, cyclizine, meclozine, buclizine.

   * Children with a history of drug hypersensitivity.
   * Pregnant, lactating or possibly pregnant female children.
   * Children with complications that may be clinically significant (e.g., hepatic disorder, renal disorder, heart disease or others) because of which they are judged as inappropriate for this trial.
   * Children who are sensitive to pollen as a duplicate allergen and whose treatment periods are thought in the pollen dispersion periods.
   * Children with vasomotor rhinitis and eosinophilic rhinitis.
   * Children complicated with a nasal disorder (e.g., acute or chronic rhinitis, hypertrophic rhinitis, acute or chronic sinusitis, deviation of nasal septum, nasal polyp, etc.) with a degree that may influence on the evaluation of the study drugs.
   * Children complicated with asthma that requires the treatment with adrenocortical hormone (including the preparations compounded with adrenocortical hormone).
   * Children administered the following drugs within one week (6days) or 4 weeks (27days) before the start of the observation period [within one week] • Anti-histamine drugs (oral, injection, and nasal drop) • Chemical mediator release inhibitors (mast cell stabilizer) • Th2 cytokine inhibitors (suplatast tosilate) • Leukotriene receptor antagonists • Thromboxane A2 receptor antagonists

     • Thromboxane synthetase inhibitors

     • Biological preparations and vaccines indicated against allergic rhinitis

     • Vasoconstrictor(oral and nasal drop)

     • Anticholinergic drugs (inhalant only)

     • General cold remedies (including OTC)

     • Herb medicines that have antiallergic action (SHOSEIRYUTO, SHOSAIKOTO, SAIBOKUTO, etc.)

     • OTC anti-rhinitis drugs (oral, inhalant, nasal drop) [within 4 weeks]

     • Adrenocortical hormones (oral [including combination drugs], injection, inhalant, nasal drop, suppository)

     • Histamine added γ-globulin preparations
   * Children who have started specific desensitization treatment or nonspecific modulation treatment but who have not reached the maintenance level of treatment.
   * Children who have received surgical treatment for reduction and modulation of nasal mucosa, redintegration therapy of nasal cavity to improve the degree of nasal airway, or surgical operation to improve rhinorrhea.
   * Children who have previously taken the investigational products of this trial.
   * Children who have participated in other clinical trial within 6 months of the date of informed consent for this clinical study or children who are participating in another trial as of the date of informed consent for this trial.
   * Children judged by the investigator or sub-investigator as inappropriate to participate in the trial.

[Before the start of treatment period] - Children whose severity score calculated by the following formula on the basis of nasal symptom score (sneezing, rhinorrhea, nasal pruritus and nasal congestion) in the baseline assessment period (3 days from D5 to D7) is 10 or higher Severity of TNSS = [TDNSS(D-3)+TDNSS(D-2)+TDNSS(D-1)]/3

* Children who have used prohibited concomitant drugs during the observation period.
* Children who have complicated acute upper airway inflammation during the observation period.
* Children who are applicable to the exclusion criteria as to the status [before the start of observation period] during the observation period." gher

Exclusion criteria:

"[Before the start of observation period]

1. Children with a history of hypersensitivity to an ingredient of cetirizine hydrochloride preparation, or hydroxyzine, cyclizine, meclozine, buclizine.
2. Children with a history of drug hypersensitivity.
3. Pregnant, lactating or possibly pregnant female children.
4. Children with complications that may be clinically significant (e.g., hepatic disorder, renal disorder, heart disease or others) because of which they are judged as inappropriate for this trial.
5. Children who are sensitive to pollen as a duplicate allergen and whose treatment periods are thought in the pollen dispersion periods.
6. Children with vasomotor rhinitis and eosinophilic rhinitis.
7. Children complicated with a nasal disorder (e.g., acute or chronic rhinitis, hypertrophic rhinitis, acute or chronic sinusitis, deviation of nasal septum, nasal polyp, etc.) with a degree that may influence on the evaluation of the study drugs.
8. Children complicated with asthma that requires the treatment with adrenocortical hormone (including the preparations compounded with adrenocortical hormone).
9. Children administered the following drugs within one week (6days) or 4 weeks (27days) before the start of the observation period [within one week]

   • Anti-histamine drugs (oral, injection, and nasal drop)

   • Chemical mediator release inhibitors (mast cell stabilizer)

   • Th2 cytokine inhibitors (suplatast tosilate)

   • Leukotriene receptor antagonists

   • Thromboxane A2 receptor antagonists

   • Thromboxane synthetase inhibitors

   • Biological preparations and vaccines indicated against allergic rhinitis

   • Vasoconstrictor(oral and nasal drop)

   • Anticholinergic drugs (inhalant only)

   • General cold remedies (including OTC)

   • Herb medicines that have antiallergic action (SHOSEIRYUTO, SHOSAIKOTO, SAIBOKUTO, etc.)
   * OTC anti-rhinitis drugs (oral, inhalant, nasal drop) [within 4 weeks]
   * Adrenocortical hormones (oral [including combination drugs], injection, inhalant, nasal drop, suppository)
   * Histamine added γ-globulin preparations
10. Children who have started specific desensitization treatment or nonspecific modulation treatment but who have not reached the maintenance level of treatment.
11. Children who have received surgical treatment for reduction and modulation of nasal mucosa, redintegration therapy of nasal cavity to improve the degree of nasal airway, or surgical operation to improve rhinorrhea.
12. Children who have previously taken the investigational products of this trial.
13. Children who have participated in other clinical trial within 6 months of the date of informed consent for this clinical study or children who are participating in another trial as of the date of informed consent for this trial.
14. Children judged by the investigator or sub-investigator as inappropriate to participate in the trial.

[Before the start of treatment period]

1） Children whose severity score calculated by the following formula on the basis of nasal symptom score (sneezing, rhinorrhea, nasal pruritus and nasal congestion) in the baseline assessment period (3 days from D5 to D7) is 10 or higher Severity of TNSS = [TDNSS(D-3)+TDNSS(D-2)+TDNSS(D-1)]/3 2) Children who have used prohibited concomitant drugs during the observation period.

3) Children who have complicated acute upper airway inflammation during the observation period.

4) Children who are applicable to the exclusion criteria as to the status [before the start of observation period] during the observation period."

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2007-07-27 (Actual); Primary Completion 2007-10-03 (Actual); Study Completion 2007-10-03 (Actual)

PRIMARY OUTCOMES:
Change in the total nasal symptom score (TNSS) during the total treatment period from the baseline | From Baseline to Day 14
  TNSS is a sum of the nasal symptom score for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The Baseline value is defined as the average TNSS over the last 3 consecutive days prior to Day 1. For total treatment period, the average TNSS for each participant was calculated using available diary data from the total treatment period, taking the average of non-missing data during the period. Change from Baseline was calculated as the score at Baseline minus the mean score for the total treatment period.

SECONDARY OUTCOMES:
Changes in TNSS on the first and the second weeks of the treatment period from the baseline | From Baseline to Day 7 and Day 14
  TNSS is a sum of the nasal symptom score for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The Baseline value is defined as the average TNSS over the last 3 consecutive days prior to Day 1. For total treatment period, the average TNSS for each participant was calculated using available diary data from the total treatment period, taking the average of non-missing data during the period. Change from Baseline was calculated as the score at Baseline minus the mean score at Week 1 and Week 2.
Mean scores for each nasal symptom and the time-course changes for the scores | From Baseline to Day 14
  Each nasal symptom score for sneezing, rhinorrhea, nasal congestion and nasal itching is scored on a scale from 0 to 3; the larger score indicates more severe symptoms. The parent/guardian or the participant scored nasal symptoms every day.
Time-course changes in a total of daily mean nasal symptom scores (TDNSS) | From Baseline to Day 14
  TDNSS is a sum of the daily nasal symptom score for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is score on a scale from 0 to 3; the range of sums for TDNSS is 0 to 12; a larger score indicates more severe symptoms.
Investigator global improvement rating on the first day of Treatment Week 2 (Day 8) and the final observation day (Day 15 ) or at discontinuation (DC) | Day 8 and Day 15 or DC
  The investigator evaluated the participant's improvement rating (defined as improvement in the symptoms of rhinitis compared with Baseline), using the following 5 categories: significantly improved, moderately improved, mildly improved, unchanged, and worsened.
Participant global improvement rating on the first day of Treatment Week 2 (Day 8) and the final observation day (Day 15) or at DC | Day 8 and Day 15 or DC
  The participant's parent/guardian or the participant evaluated the participant's improvement rating (defined as improvement in the symptoms of rhinitis compared with Baseline), using the following 7 categories: significantly improved, improved, slightly improved, unchanged, slightly worsened, worsened, and significantly worsened.
Changes in each rhinoscopy finding (swelling and color of inferior conchal mucosa and aqueous secretion volume (ASV)) on first day of Treatment Week 1 (Day 1), the first day of Treatment Week 2 (Day 8) and the final observation day (Day 15) or at DC | Day 1, Day 8 and Day 15 or DC
  Rhinoscopy was assessed by the investigator by scoring swelling of inferior conchal mucosa scored as 0 (none), 1 (possible to see center of the middle turbinate), 2 (between 1 and 3), or 3 (impossible to see middle turbinate); color of inferior conchal mucosa scored as 0 (normal), 1 (pink), 2 (red), or 3 (pale); aqueous secretion volume (vol) scored as 0 (none), 1 (small amount adhered), 2 (between 1 and 3), or 3 (filled).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo